CLINICAL TRIAL: NCT00081965
Title: Acupuncture for the Treatment of Hot Flashes in Breast Cancer Patients: A Randomized Controlled Trial
Brief Title: Acupuncture in Treating Hot Flashes in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: 02-108; MSKCC-02108A
Record Dates: First submitted 2004-04-27; First posted 2004-04-28 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer; Hot Flashes
Keywords: breast cancer in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IV breast cancer; recurrent breast cancer; stage IIIC breast cancer; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes; Breast Carcinoma In Situ | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: acupuncture therapy
Procedure: hot flashes attenuation
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Acupuncture may help relieve hot flashes in women with breast cancer. It is not yet known whether acupuncture is more effective than a placebo in treating hot flashes in women with breast cancer

PURPOSE: This randomized clinical trial is studying acupuncture to see how well it works compared to a placebo in treating hot flashes in women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether acupuncture, compared to placebo, reduces the incidence of hot flashes in women with breast cancer.

Secondary

* Determine the long-term effects of acupuncture on hot flashes.

OUTLINE: This a randomized, placebo-controlled, multicenter study. Patients are stratified according to concurrent treatment with selective estrogen receptor modulators, gonadotropin-releasing hormone analogs, or aromatase inhibitors (yes vs no), concurrent use of hot flash medication or selective serotonin reuptake inhibitors (SSRIs) (yes vs no), baseline hot flash frequency (> 7 per day), and menopausal status at diagnosis (premenopausal vs postmenopausal). Patients are randomized to 1 of 2 treatment arms.

* Arm I (treatment): Patients receive 8 acupuncture treatments over 4 weeks.
* Arm II (control): Patients receive 8 placebo acupuncture treatments over 4 weeks. Beginning at week 7, patients are offered 8 true acupuncture treatments over 4 weeks.

Patients in both arms complete a "hot flash" diary for 1 week before treatment and then periodically during and after treatment.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer (including in situ disease)
* Must be receiving treatment for breast cancer at Memorial Sloan Kettering Cancer Center (MSKCC) or its regional site (Commack)
* Has an average of 3 or more hot flashes a day during 1 week of baseline diary recording
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Pre- or postmenopausal
* Karnofsky performance status 70-100%
* Ambulatory
* No skin infection

PRIOR CONCURRENT THERAPY:

* More than 3 weeks since prior and no concurrent treatment with any of the following during the 6 week evaluation period of the trial:

  * Surgery
  * Initiation of a new chemotherapy regimen
  * Initiation of immunotherapy
  * Initiation of radiotherapy
  * Initiation or cessation of hormonal therapy
* More than 6 weeks since prior acupuncture treatment (6 months for acupuncture specifically for the treatment of hot flashes)
* No concurrent pharmacological treatment for hot flashes unless dose has been stable for 4 weeks
* No concurrent selective serotonin reuptake inhibitors (SSRIs) unless dose has been stable for 4 weeks

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of hot flashes, as measured by a hot flash diary

CONTACTS AND LOCATIONS:
Overall Officials: Barrie R. Cassileth, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Deng G, Vickers A, Yeung S, D'Andrea GM, Xiao H, Heerdt AS, Sugarman S, Troso-Sandoval T, Seidman AD, Hudis CA, Cassileth B. Randomized, controlled trial of acupuncture for the treatment of hot flashes in breast cancer patients. J Clin Oncol. 2007 Dec 10;25(35):5584-90. doi: 10.1200/JCO.2007.12.0774. PMID 18065731